CLINICAL TRIAL: NCT05499468
Title: Evaluating a Physician Popular Opinion Leader-Led Intervention to Encourage Postgraduate Trainee Participation in One-On-One Support Resources
Brief Title: Evaluating a Physician Opinion Leader Intervention to Increase Utilization of Coaching/Therapy During Residency
Acronym: POL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: The Physicians Foundation (Unknown)
Responsible Party: Principal Investigator, Mickey Trockel, Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 60993
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Workplace Culture; Help-Seeking Behavior; Social Stigma; Education, Medical, Continuing
Keywords: Occupational Culture; Trainee Mental Health; Physician Stigma; Resident Health Promotion
MeSH Terms: conditions — Help-Seeking Behavior; Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Popular-Opinion Leader-led workshops & conversations to encourage utilization of support resources (Other): Physicians identified by programwide Qualtrics survey item asking housestaff who in their program they respect and trust most, personally and professionally. Identified POLs were invited to join this health promotion effort as a POL to improve the culture of wellness and psychological safety among housestaff and encourage them to utilize resources at a time when they may benefit significantly. POLs were trained to endorse the benefits of mental health promotion coaching or therapy for residents training at Stanford.
  Interventions: Other: Popular-Opinion Leader-led encouragement during training meetings and informal conversation
- Standard Training Program Curriculum and Access to Existing Support Resources (No Intervention): All residents and fellows continued to have the same access to coaching and psychotherapy resources available through Stanford WellConnect, along with other educational activities in their usual training.

INTERVENTIONS:
Other: Popular-Opinion Leader-led encouragement during training meetings and informal conversation — Investigators adapted evidence-based principles from the Popular Opinion Leader framework to increase utilizations of existing one-on-one emotional support resources for physicians-in-training at Stanford (an effective HIV prevention intervention developed by the CDC for changing social norms and reducing behavioral risk factors led by influential members of a community, trained to promote behavior change). All intervention activities designed to encourage utilization were delivered as part of health promotion during pre-existing clinical training meetings and no data was collected during these workshops. Identified POLs were recruited and trained to encourage their colleagues to use existing support resources and engage in two 30-60 minute workshops scheduled to occur during training meetings.
  Arms: Popular-Opinion Leader-led workshops & conversations to encourage utilization of support resources

SUMMARY:
Investigators will assess the efficacy of a physician popular opinion leader-led intervention to increase awareness and utilization of existing evidence-based coaching or therapy among post-graduate clinical trainees at Stanford.

DETAILED DESCRIPTION:
All Stanford residents are provided access to evidence-based coaching and/or therapy, such as cognitive and behavioral targeting of drivers of burnout.

The present project evaluates the ability of a popular opinion leader approach to normalize use of these resources with the hope of increasing utilization. Over the ark of 31 months, all training programs will receive the intervention.

A flexible, minimally intrusive, residency-randomized cluster design will be used to determine the sequence of which programs receive the intervention immediately verses delayed. Investigators delivered an intervention adapted from the CDC Popular Opinion Leader framework for encouraging physicians to utilize existing resources for individual support during residency through Stanford WellConnect (a confidential mental health promotion program for medical residents, fellows, and all benefits-eligible faculty in the School of Medicine at Stanford during their training). Support resources include evidence-based coaching and/or therapy, such as cognitive and behavioral targeting of drivers of burnout for which physicians are at higher-than-average risk. All health promotion efforts were delivered as part of clinical training, outside the scope of this distinct research evaluation. No data has been collected from individual POLs or workshop participants to date.

Investigators will utilize administratively collected data from postgraduate physician trainee populations across 20 Stanford paired residency programs with 5 or more house-staff (residents or fellows) each. 10 programs were randomly assigned to be the first to receive the intervention, and 10 to a delayed intervention group (10 programs). The immediate intervention arm (vs. delayed) received a POL-led health promotion intervention delivered as part of their regular postgraduate medical training educational activities (e.g., during didactic sessions), designed to encourage them to consider participating in existing, evidence-based one-on-one support resources (coaching and therapy with trained professionals) available through WellConnect. The POL intervention includes two formal workshop discussions and informal conversations with trained physician POL colleagues. The delayed intervention arm continued to receive their regular postgraduate medical training educational activities as well as access to the same coaching and therapy resources through WellConnect, and any other wellness resources involved in the curriculum at each program as the immediate intervention arm. The delayed intervention arm will also receive the POL program from November 1st 2022 through May 2023.

The investigators will evaluate multiple outcomes between the immediate and delayed intervention arms using administratively collected WellConnect usage data (% of each program who participate in coaching or therapy from each enrolled residency program population during the trial). In addition, investigators will analyze administratively collected institutional wellness survey data to determine population level differences in perceptions of stigma against mental health support, self-valuation, burnout, and professional fulfillment.

ELIGIBILITY:
Inclusion Criteria:

* This post-test only evaluation study will use de-identified data that investigators will request after administrative survey data is collected by the organization
* The primary aim dataset will include WellConnect program level usage data, indicating the total aggregate number of service requests from the cohorts of physicians in the 20 postgraduate training programs at Stanford whose program directors opted to allow their trainees to participate in the Popular Opinion Leader-led population health promotion intervention
* The data set for secondary aims will include completely de-identified data from all house-staff who are enrolled in programs participating in the POL program, and who completed the regularly scheduled institutional wellness survey

Exclusion Criteria:

* Nonphysicians
* Those outside 20 training programs cohorts participating in the POL intervention at Stanford

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
Number of participants enrolled in WellConnect program | study week 7, program usage report will be requested from WellConnect Coordinator in October 2022
  The WellConnect service tracks utilization by residents in each department. The study team will ask WellConnect to report the total number of calls from November 1, 2021, through June 30th 2022, from house-staff (residents and fellows) who are part of training programs that participated in the POL program. The proportion of residents in each program who participate in coaching or psychotherapy support offered by the WellConnect program will be calculated by dividing the number of residents who participate in the program by the total number of residents enrolled in the program.

SECONDARY OUTCOMES:
Score in "Disclosure and Help-Seeking" Subscale of the Opening Minds Stigma Scale for Health Care Providers (from administratively collected institutional wellness survey data) | study week 7, post-intervention, de-identified data will be requested from organization-wide administratively collected survey data. This data will be requested in December, 2022
  "Disclosure and Help-seeking subscale" is a subscale of the Opening Minds Scale for Health Care Providers (OMS-HC) includes 4 items, with responses on a Likert scale (scores range from 1 to 5, where a higher score is less favorable). Respondents are instructed "These questions ask you to agree or disagree with a series of statements about mental illness. There is no correct answer. Please mark the box that best fits your opinion" and statements include: 1) "If I were under treatment for a mental illness I would not disclose this to any of my colleagues"; 2) "I would see myself as weak if I had a mental illness and could not fix it myself"; 3) "I would be reluctant to seek help if I had a mental illness"; and 4) "If I had a mental illness, I would tell my friends."
Response to standardized question from the National Comorbidity Survey ("Attitudes Regarding Help Seeking" item) from administratively collected institutional wellness survey data | study week 7, post-intervention de-identified data will be requested from organization-wide administratively collected survey data. This data will be requested in December, 2022.
  Assessed using a single standardized item from the National Comorbidity Survey, which asks "People differ a lot in their feelings about professional help for emotional problems. If you had a serious emotional problem, would you definitely go for professional help, probably go, probably not go, or definitely not go for professional help?" Responses (ranging from most to least favorable) are: "Would definitely go," "Would probably go," "Would probably not go," and "Would definitely not go." Source: Mojtabai R, Evans-Lacko S, Schomerus G, Thornicroft G. Attitudes Toward Mental Health Help Seeking as Predictors of Future Help-Seeking Behavior and Use of Mental Health Treatments. Psychiatr Serv. 2016 Jun 1;67(6):650-7. doi: 10.1176/appi.ps.201500164. Epub 2016 Feb 14. PMID: 26876662.
Stanford Professional Fulfillment Index Score (from administratively collected institutional wellness survey data) | study week 7, post-intervention de-identified data will be requested from organization-wide administratively collected survey. This data will be requested in December, 2022.
  Each PFI item is scored from 0 to 4, using the associated five-point Likert scale. Scale scores are then calculated by averaging the items scores of all item within each corresponding scale, such that all scale scores also range from 0 to 4, which are then converted to a scale of 0-10.
  Using 0-10 scale, the cut-point for Professional fulfillment is 7.5 and greater (higher score more favorable, and for Overall Burnout is 3.325 and greater (lower score more favorable). Professional fulfillment scale cut-point is 7.5. Those with average scores of 7.5 and greater are more likely to be professionally fulfilled. Overall Burnout, has a cut-point of 3.325. Those with averages scores of 3.325 or greater are more likely to be experiencing Burnout.
Self-Valuation Index Score (from administratively collected institutional wellness survey data) | study week 7, post-intervention de-identified data will be requested from organization-wide administratively collected survey data. This data will be requested in December, 2022
  Self-valuation is a construct "involving constructive prioritization of personal well-being and a growth mindset perspective that seeks to learn and improve as the primary response to errors," assessed using 4-item questionnaire that asks respondents to characterize their experiences in the past 2 weeks, measured using "a 5-point (0-4) Likert scale (summative score range, 0-16, higher score more favorable)," where total self valuation index score is calculated by adding up individual item scores.

CONTACTS AND LOCATIONS:
Overall Officials: Mickey T Trockel, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kassam A, Papish A, Modgill G, Patten S. The development and psychometric properties of a new scale to measure mental illness related stigma by health care providers: the Opening Minds Scale for Health Care Providers (OMS-HC). BMC Psychiatry. 2012 Jun 13;12:62. doi: 10.1186/1471-244X-12-62. PMID 22694771
- [Background] Trockel M, Bohman B, Lesure E, Hamidi MS, Welle D, Roberts L, Shanafelt T. A Brief Instrument to Assess Both Burnout and Professional Fulfillment in Physicians: Reliability and Validity, Including Correlation with Self-Reported Medical Errors, in a Sample of Resident and Practicing Physicians. Acad Psychiatry. 2018 Feb;42(1):11-24. doi: 10.1007/s40596-017-0849-3. Epub 2017 Dec 1. PMID 29196982
- [Background] Trockel MT, Hamidi MS, Menon NK, Rowe SG, Dudley JC, Stewart MT, Geisler CZ, Bohman BD, Shanafelt TD. Self-valuation: Attending to the Most Important Instrument in the Practice of Medicine. Mayo Clin Proc. 2019 Oct;94(10):2022-2031. doi: 10.1016/j.mayocp.2019.04.040. Epub 2019 Sep 19. PMID 31543254
- [Background] NIMH Collaborative HIV/STD Prevention Trial Group. The community popular opinion leader HIV prevention programme: conceptual basis and intervention procedures. AIDS. 2007 Apr;21 Suppl 2:S59-68. doi: 10.1097/01.aids.0000266458.49138.fa. PMID 17413265
- [Background] Shanafelt TD, Dyrbye LN, West CP, Sinsky C, Tutty M, Carlasare LE, Wang H, Trockel M. Suicidal Ideation and Attitudes Regarding Help Seeking in US Physicians Relative to the US Working Population. Mayo Clin Proc. 2021 Aug;96(8):2067-2080. doi: 10.1016/j.mayocp.2021.01.033. Epub 2021 Jul 20. PMID 34301399
- [Background] Mojtabai R, Evans-Lacko S, Schomerus G, Thornicroft G. Attitudes Toward Mental Health Help Seeking as Predictors of Future Help-Seeking Behavior and Use of Mental Health Treatments. Psychiatr Serv. 2016 Jun 1;67(6):650-7. doi: 10.1176/appi.ps.201500164. Epub 2016 Feb 14. PMID 26876662